CLINICAL TRIAL: NCT03172676
Title: Effects of Helicobacter Pylori Eradication Therapy in Children With Chronic Immune Thrombocytopenic Purpura
Brief Title: Effects of Helicobacter Pylori Eradication in Children With Chronic Immune Thrombocytopenic Purpura
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mary Makram Kamel, principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITPHP
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Amoxicillin; Clarithromycin; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Helicobacter pylori negative patients (No Intervention): chronic immune thrombocytopenic purpura patients who will be diagnosed negative for Helicobacter pylori infection using detection of Helicobacter pylori antigen in stool of these patients.
- Helicobacter pylori positive patients with intervention (Active Comparator): chronic immune thrombocytopenic purpura patients who will be diagnosed positive for Helicobacter pylori infection using detection of Helicobacter pylori antigen in stool of these patients will receive treatment of Helicobacter pylori: Amoxicillin for 14 days, Clarithromycin for 14 days and Proton pump inhibitor for one month).
  Interventions: Drug: Amoxicillin 50 mg/kg/day in 2 divided doses for 14 days.; Drug: Clarithromycin 15 mg/kg/day in 2 divided doses for 14 days.; Drug: Proton pump inhibitor 1 mg/kg/day in 2 divided doses 1 month
- Helicobacter pylori positive patients without intervention (No Intervention): chronic immune thrombocytopenic purpura patients who will be diagnosed positive for Helicobacter pylori infection using detection of Helicobacter pylori antigen in stool of these patients will not receive treatment of Helicobacter pylori during the study,these patient group will receive treatment of Helicobacter pylori after the end of the study

INTERVENTIONS:
Drug: Amoxicillin 50 mg/kg/day in 2 divided doses for 14 days. — chronic immune thrombocytopenic purpura patients who will be diagnosed positive for helicobacter pylori infection will receive Amoxicillin for 14 days.
  Arms: Helicobacter pylori positive patients with intervention
Drug: Clarithromycin 15 mg/kg/day in 2 divided doses for 14 days. — chronic immune thrombocytopenic purpura patients who will be diagnosed positive for helicobacter pylori infection will receive Clarithromycin for 14 days.
  Arms: Helicobacter pylori positive patients with intervention
Drug: Proton pump inhibitor 1 mg/kg/day in 2 divided doses 1 month — chronic immune thrombocytopenic purpura patients who will be diagnosed positive for helicobacter pylori infection will receive proton pump inhibitor for 1 month.
  Arms: Helicobacter pylori positive patients with intervention

SUMMARY:
Thrombocytopenia refers to a reduction in platelet count to (<150 × 109/L). Immune thrombocytopenic purpura is an acquired autoimmune disorder defined by isolated thrombocytopenia and the exclusion of other causes of thrombocytopenia

DETAILED DESCRIPTION:
Helicobacter pylori was recently demonstrated as an etiological factor in immune thrombocytopenic purpura in some prospective studies, with reports of platelet numbers increasing in these patients after Helicobacter pylori eradication treatment.However, other studies have shown a negative result after eradication treatment of Helicobacter pylori infection in patients with chronic immune thrombocytopenic purpura, leading to controversy.

ELIGIBILITY:
Inclusion Criteria:

1. chronic immune thrombocytopenic purpura patients who still have thrombocytopenia > 12 months
2. age <18 years .
3. diagnosis of immune thrombocytopenic purpura according to American Society of Hematology criteria based on an initial platelet count <100×103/μL .
4. Patients diagnosed as steroid and immunoglobulin resistant chronic immune thrombocytopenic purpura .

exclusion criteria:

1. Patients with acute immune thrombocytopenic purpura . .
2. age >18 years.
3. thrombocytopenia was related to autoimmune disorders, drugs, a family history consistent with inherited thrombocytopenia, human immunodeficiency virus infection, hepatitis.
4. previous history of Helicobacter pylori eradication; and history of medication with proton pump inhibitors, H2- receptor antagonists, or antibiotics in the previous 4 weeks.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
effects of Helicobacter pylori infection eradication on platelet counts of chronic immune thrombocytopenic patients | 6 months
  platelet counts will be measured at the start of the study ,before the starting of the interventions, and after 6 months. platelet response will be classified as: 1-complete response: platelet count> 150 × 109/L , 2-partial response: platelet count : 50-150 × 109/L , no response: platelet count < 50 × 109/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Medical School, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loffredo G, Marzano MG, Migliorati R, Miele E, Menna F, Poggi V, Staiano A. The relationship between immune thrombocytopenic purpura and Helicobacter pylori infection in children: where is the truth? Eur J Pediatr. 2007 Oct;166(10):1067-8. doi: 10.1007/s00431-006-0344-4. Epub 2006 Nov 29. No abstract available. PMID 17136353
- [Background] Chey WD, Leontiadis GI, Howden CW, Moss SF. ACG Clinical Guideline: Treatment of Helicobacter pylori Infection. Am J Gastroenterol. 2017 Feb;112(2):212-239. doi: 10.1038/ajg.2016.563. Epub 2017 Jan 10. PMID 28071659
- [Background] Treepongkaruna S, Sirachainan N, Kanjanapongkul S, Winaichatsak A, Sirithorn S, Sumritsopak R, Chuansumrit A. Absence of platelet recovery following Helicobacter pylori eradication in childhood chronic idiopathic thrombocytopenic purpura: a multi-center randomized controlled trial. Pediatr Blood Cancer. 2009 Jul;53(1):72-7. doi: 10.1002/pbc.21991. PMID 19301380